CLINICAL TRIAL: NCT02078271
Title: Food-Based Intervention and Psychosocial Stimulation to Improve Growth & Development of < 24 Month Indonesian Children
Acronym: FIRST
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Indonesia University (Other)
Collaborators: Nestlé Foundation (Other)
Responsible Party: Principal Investigator, Umi Fahmida, PhD, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: FIRST
Record Dates: First submitted 2014-02-24; First posted 2014-03-05 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Nutritional Anemia; Child Development
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- FBDG group (Experimental): The group received Food Based Dietary Guidelines for feeding recommendation. Monthly-session with group of mothers involving interactive activities e.g. cooking session, cooking competition and games.
  Interventions: Other: FBDG group
- Stimulation group (Experimental): The children received psychosocial stimulation from the mothers. Mothers were taught on psychosocial module which was developed using locally existing resources and was directed at improving four aspects of child development, namely gross motoric, fine motor, language and socio-emotional developments.
  Interventions: Other: Stimulation
- Combined (FBDG and Stimulation) (Experimental): The group received both FBDG and psychosocial stimulation
  Interventions: Other: FBDG group; Other: Stimulation; Other: Combinded FBDG and stimulation
- Control (Other): The group received standard health education messages from existing health care system.
  Interventions: Other: Control group

INTERVENTIONS:
Other: FBDG group — The group received food based dietary guidelines for complementary feeding
  Other Names: Food Based Dietary Guidelines
  Arms: Combined (FBDG and Stimulation); FBDG group
Other: Stimulation — The group received psychosocial stimulation
  Arms: Combined (FBDG and Stimulation); Stimulation group
Other: Combinded FBDG and stimulation — The group received both FBDG and psychosocial stimulation
  Arms: Combined (FBDG and Stimulation)
Other: Control group
  Arms: Control

SUMMARY:
WHO has urged all developing countries to develop programmes to improve complementary-feeding (CF) practices because of their importance for optimal growth, development and health of infants and young children While supplementation programmes and/or highly-fortified "super-foods" have limited success in improving CF-practices in disadvantaged environments, population-specific food-based dietary guidelines (FBDG), based on locally-available foods and requires minimal changes to local food pattern, will enhance the chances of programme success.

Our previous study was able to identify the need for, potential and finally develop FBDG for CF of 6-8mo and 9-11mo infants using combined linear-and-goal programming approach (LP approach). This research is therefore being made to support the next phase of the study i.e. to assess the efficacy of FBDG, for improving CF/dietary-practices and growth in <24mo children (window of opportunity). As growth and development is inter-related, home-based stimulation will be included in this trial to see the effect on child development. While studies have shown that stimulation at early age benefits children through their late adolescence; evidence from Indonesia is lacking. This study therefore aims to see the effect on growth and development of community trial using food-based dietary guideline and stimulation. It is expected that findings from this study will provide scientific evidence as the basis for program formulation.

ELIGIBILITY:
Inclusion Criteria:

* children aged 9-11 month on enrolment,
* weight-for-age Z-score <-1.00 but >-3.00

Exclusion Criteria:

* having mental or physical disabilities

Ages: 9 Months to 11 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 480 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Nutritional status | baseline (before intervention), endline (6 months after intervention), and follow up (2 years after endline)
  Anthropometry status (Height for age, weight for height, weight for age, BMI for age), Hemoglobin, iron status (serum ferritin, transferrin receptor), vitamin A status (RBP). Iron and vitamin A status were measured only at follow up
Child development | baseline (before intervention), endline (6 months after intervention), and follow up (2 years after endline)
  Child development was measured using Bayley Scale of Infant Development II (BSID-II) at baseline and 6mo after the intervention (endline). Two years after the endline (the follow-up), child development was measured using Wechsler Preschool and Primary Scale of Intelligence - Fourth Edition (WPPSI-IV).

CONTACTS AND LOCATIONS:
Overall Officials: Umi Fahmida, PhD, Principal Investigator — SEAMEO-RECFON, University of Indonesia
Locations (1):
- South East Asian Ministers of Education Organization, Regional Center for Food and Nutrition (SEAMEO-RECFON), Jakarta, Java, Indonesia

REFERENCES:
- [Background] Adu-Afarwuah S, Lartey A, Brown KH, Zlotkin S, Briend A, Dewey KG. Home fortification of complementary foods with micronutrient supplements is well accepted and has positive effects on infant iron status in Ghana. Am J Clin Nutr. 2008 Apr;87(4):929-38. doi: 10.1093/ajcn/87.4.929. PMID 18400716
- [Background] Bradley RH, Corwyn RF, McAdoo HP, Coll CG. The home environments of children in the United States part I: variations by age, ethnicity, and poverty status. Child Dev. 2001 Nov-Dec;72(6):1844-67. doi: 10.1111/1467-8624.t01-1-00382. PMID 11768149
- [Background] Engle PL, Zeitlin M. Active feeding behavior compensates for low interest in food among young Nicaraguan children. J Nutr. 1996 Jul;126(7):1808-16. doi: 10.1093/jn/126.7.1808. PMID 8683342
- [Background] Ferguson EL, Darmon N, Briend A, Premachandra IM. Food-based dietary guidelines can be developed and tested using linear programming analysis. J Nutr. 2004 Apr;134(4):951-7. doi: 10.1093/jn/134.4.951. PMID 15051853
- [Background] Ferguson EL, Darmon N, Fahmida U, Fitriyanti S, Harper TB, Premachandra IM. Design of optimal food-based complementary feeding recommendations and identification of key "problem nutrients" using goal programming. J Nutr. 2006 Sep;136(9):2399-404. doi: 10.1093/jn/136.9.2399. PMID 16920861
- [Background] Hamadani JD, Huda SN, Khatun F, Grantham-McGregor SM. Psychosocial stimulation improves the development of undernourished children in rural Bangladesh. J Nutr. 2006 Oct;136(10):2645-52. doi: 10.1093/jn/136.10.2645. PMID 16988140
- [Background] Gardner JM, Powell CA, Baker-Henningham H, Walker SP, Cole TJ, Grantham-McGregor SM. Zinc supplementation and psychosocial stimulation: effects on the development of undernourished Jamaican children. Am J Clin Nutr. 2005 Aug;82(2):399-405. doi: 10.1093/ajcn.82.2.399. PMID 16087985
- [Background] Santika O, Fahmida U, Ferguson EL. Development of food-based complementary feeding recommendations for 9- to 11-month-old peri-urban Indonesian infants using linear programming. J Nutr. 2009 Jan;139(1):135-41. doi: 10.3945/jn.108.092270. Epub 2008 Dec 3. PMID 19056658
- [Background] Walker SP, Chang SM, Powell CA, Grantham-McGregor SM. Effects of early childhood psychosocial stimulation and nutritional supplementation on cognition and education in growth-stunted Jamaican children: prospective cohort study. Lancet. 2005 Nov 19;366(9499):1804-7. doi: 10.1016/S0140-6736(05)67574-5. PMID 16298218
- [Background] Walker SP, Chang SM, Powell CA, Simonoff E, Grantham-McGregor SM. Effects of psychosocial stimulation and dietary supplementation in early childhood on psychosocial functioning in late adolescence: follow-up of randomised controlled trial. BMJ. 2006 Sep 2;333(7566):472. doi: 10.1136/bmj.38897.555208.2F. Epub 2006 Jul 28. PMID 16877454
- [Background] Walker SP, Chang SM, Powell CA, Simonoff E, Grantham-McGregor SM. Early childhood stunting is associated with poor psychological functioning in late adolescence and effects are reduced by psychosocial stimulation. J Nutr. 2007 Nov;137(11):2464-9. doi: 10.1093/jn/137.11.2464. PMID 17951486
- [Derived] Fahmida U, Kolopaking R, Santika O, Sriani S, Umar J, Htet MK, Ferguson E. Effectiveness in improving knowledge, practices, and intakes of "key problem nutrients" of a complementary feeding intervention developed by using linear programming: experience in Lombok, Indonesia. Am J Clin Nutr. 2015 Mar;101(3):455-61. doi: 10.3945/ajcn.114.087775. Epub 2014 Dec 24. PMID 25733629